CLINICAL TRIAL: NCT04023071
Title: A Phase I Study of FT516 as Monotherapy in Relapsed/Refractory Acute Myelogenous Leukemia and in Combination With Monoclonal Antibodies in Relapsed/Refractory B-Cell Lymphoma
Brief Title: FT516 in Subjects With Advanced Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor.
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT516-101
Record Dates: First submitted 2019-07-09; First posted 2019-07-17 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acute Myelogenous Leukemia; B-cell Lymphoma
Keywords: AML; Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, B-Cell; Lymphoma | interventions — Rituximab; obinutuzumab; Cyclophosphamide; fludarabine; Interleukin-2; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FT516 Monotherapy (Experimental): FT516 monotherapy in adult subjects with r/r AML.
  Interventions: Drug: FT516; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2
- FT516 in Combination with Monoclonal Antibodies (Experimental): FT516 in combination with one of the following monoclonal antibodies in adult subjects with r/r B-cell lymphoma: rituximab or obinutuzumab.
  Interventions: Drug: FT516; Drug: Rituximab; Drug: Obinutuzumab; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2
- FT516 in Combination with Monoclonal Antibodies on an Extended-Dosing Schedule (Experimental): FT516 on an extended-dosing schedule in combination with one of the following monoclonal antibodies in adult subjects with r/r B-cell lymphoma: rituximab or obinutuzumab.
  Interventions: Drug: FT516; Drug: Rituximab; Drug: Obinutuzumab; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2
- FT516 in Combination with Monoclonal Antibodies following Bendamustine Conditioning (Experimental): Bendamustine conditioning followed by FT516 in combination with one of the following monoclonal antibodies in adult subjects with r/r B-cell lymphoma: rituximab or obinutuzumab.
  Interventions: Drug: FT516; Drug: Rituximab; Drug: Obinutuzumab; Drug: IL-2; Drug: Bendamustine

INTERVENTIONS:
Drug: FT516 — Experimental Interventional Therapy
Drug: Rituximab — Monoclonal Antibody
  Other Names: Rituxan; MabThera
  Arms: FT516 in Combination with Monoclonal Antibodies; FT516 in Combination with Monoclonal Antibodies following Bendamustine Conditioning; FT516 in Combination with Monoclonal Antibodies on an Extended-Dosing Schedule
Drug: Obinutuzumab — Monoclonal Antibody
  Other Names: Gazyva
  Arms: FT516 in Combination with Monoclonal Antibodies; FT516 in Combination with Monoclonal Antibodies following Bendamustine Conditioning; FT516 in Combination with Monoclonal Antibodies on an Extended-Dosing Schedule
Drug: Cyclophosphamide — Conditioning agent
  Arms: FT516 Monotherapy; FT516 in Combination with Monoclonal Antibodies; FT516 in Combination with Monoclonal Antibodies on an Extended-Dosing Schedule
Drug: Fludarabine — Conditioning agent
  Arms: FT516 Monotherapy; FT516 in Combination with Monoclonal Antibodies; FT516 in Combination with Monoclonal Antibodies on an Extended-Dosing Schedule
Drug: IL-2 — Biologic response modifier
Drug: Bendamustine — Conditioning agent
  Other Names: Bendeka; Treanda
  Arms: FT516 in Combination with Monoclonal Antibodies following Bendamustine Conditioning

SUMMARY:
This is a Phase 1/1b dose-finding study of FT516 as monotherapy in acute myeloid leukemia (AML) and in combination with CD20 directed monoclonal antibodies in B-cell lymphoma. The study includes three stages: dose escalation, safety confirmation, and dose expansion.

ELIGIBILITY:
KEY INCLUSION CRITERIA:

Diagnosis of the following:

Regimen A (FT516 monotherapy):

* Primary Refractory AML
* Relapsed AML defined as not in CR after 1 or more re-induction attempts; if >60 years of age, prior re-induction therapy is not required

Regimen B (FT516 + rituximab or obinutuzumab):

* Histologically documented B-cell lymphoma expected to express CD20 who have relapsed after or failed to respond to at least on prior treatment regimen and for whom there is no available therapy expected to improve survival.

All subjects:

* Provision of signed and dated informed consent form (ICF)
* Age ≥18 years old
* Stated willingness to comply with study procedures and duration
* Presence of measurable disease

KEY EXCLUSION CRITERIA:

All subjects:

* Females of reproductive potential who are pregnant or lactating, and males or females not willing to use a highly effective form of contraception from Screening through the end of the study
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥2
* Evidence of insufficient organ function
* Receipt of therapy within 2 weeks prior to Cycle 1 Day 1 or within five half-lives, whichever is shorter; or any investigational therapy within 28 days prior to Cycle 1 Day 1
* Currently receiving or likely to require systemic immunosuppressive therapy
* Prior allogeneic HSCT or allogeneic CAR-T within 6 months of Cycle 1 Day 1, or ongoing requirement for systemic graft-versus-host therapy
* Receipt of an allograft organ transplant
* Known active central nervous system (CNS) involvement by malignancy.
* Clinically significant cardiovascular disease
* Clinically significant infections including: Known HIV infection; Known active Hepatitis B (HBV) or Hepatitis C (HCV) infection
* Live vaccine <6 weeks prior to start of lympho-conditioning
* Known allergy to human albumin and DMSO

Additional Exclusion Criteria for FT516 monotherapy Regimen: Diagnosis of promyelocytic leukemia with t(15:17) translocation

Additional Exclusion Criteria for FT516 plus monoclonal antibody Regimens: Diagnosis of Waldenstrom macroglobulinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
The incidence of subjects with Dose Limiting Toxicities within each dose level cohort. | Day 29
Incidence, nature, and severity of AEs, of FT516 as monotherapy in r/r AML and in combination with rituximab or obinutuzumab in r/r B-cell lymphoma. | Up to 5 years

SECONDARY OUTCOMES:
Investigator-assessed anti-tumor activity of FT516 as monotherapy in r/r AML and in combination with rituximab or obinutuzumab in r/r B-cell lymphoma. | Cycle 2 Day 29
FT516 pharmacokinetic data | Cycle 1 and Cycle 2 Study Days: 1, 2, 4, 8, 11, 15, 18, 22, 29, and Cycle 2 Day 43 and Cycle 2 Day 57.
  Percentage of donor DNA measured at each timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics
Locations (7):
- United States (7):
  - Mayo Clinic, Phoenix, Arizona
  - UC San Diego, San Diego, California
  - University of Colorado, Denver, Denver, Colorado
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - UT Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strati P, Castro J, Goodman A, Bachanova V, Kamdar M, Awan FT, Solomon SR, Wong L, Wong C, Patel D, Bickers C, Zhao W, Bashir Z, Valamehr B, Elstrom RL, Patel K. Off-the-shelf induced pluripotent stem-cell-derived natural killer-cell therapy in relapsed or refractory B-cell lymphoma: a multicentre, open-label, phase 1 study. Lancet Haematol. 2025 Jul;12(7):e505-e515. doi: 10.1016/S2352-3026(25)00142-5. PMID 40610174